CLINICAL TRIAL: NCT02476318
Title: A Study to Evaluate the Safety and Performance of ArterX™ Vascular Sealant in Sealing Synthetic Arterial Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tenaxis Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-008
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Vascular Disease
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ArterX Vascular Sealant (Experimental)
  Interventions: Device: ArterX Vascular Sealant

INTERVENTIONS:
Device: ArterX Vascular Sealant

SUMMARY:
A prospective, multi-center study to evaluate the safety and performance outcomes of the ArterX Vascular Sealant when used for prophylactic sealing of suture lines at the anastomosis between native vessel and synthetic vascular grafts.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be ≥ 18 years old
2. The subject must be scheduled for surgical placement of a synthetic graft for large vessel repair/ arterial reconstruction/ hemodialysis access.
3. The subject has no child bearing potential or has a negative serum or urine pregnancy test within 7 days of the index procedure.
4. The subject is willing and able to be contacted for minimum of 6 weeks follow up.
5. The subject or guardian must provide written informed consent using a form that is reviewed and approved by the Ethics Committee.

Exclusion Criteria:

1. The subject has a known hypersensitivity or contraindication to heparin, bovine or seafood products.
2. The subject has a history of bleeding diathesis or coagulopathy, or will refuse blood transfusion.
3. The subject is currently enrolled in this, or another investigational device or drug trail that has not completed the required follow-up period.
4. ArterX Vascular Sealant should not be used in patients who have exhibited an allergic reaction to materials of shellfish or bovine origin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Number of anastomoses with immediate sealing of the suture line | Intraoperative
  Immediate suture line sealing on clamp removal, as evidenced by a lack of clinically significant bleeding. A minimum of 50% of the anastomoses were expected to be sealed immediately.

CONTACTS AND LOCATIONS:
Overall Officials: Hans J Florek, MD, Principal Investigator — Krankenhaus Dresden Friedrichstadt Dresden, Germany
Locations (3):
- Germany (3):
  - Klinikum der Universitat zu Koln, Cologne
  - Krankenhaus Dresden Friedrichstadt, Dresden
  - Chirugische Uni Klinikum, Ulm